CLINICAL TRIAL: NCT05281055
Title: Taiwan Registry of Endovascular Thrombectomy for Acute Ischemic Stroke
Acronym: TREAT-AIS
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201708026RINA
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EVT group: Patients who received endovascular thrombectomy for acute ischemic stroke with large vessel occlusion.
  Interventions: Procedure: Endovascular thrombectomy

INTERVENTIONS:
Procedure: Endovascular thrombectomy — Timely thrombectomy for acute ischemic stroke patients with large vessel occlusion by either stent retriever, thrombosuction, others, or combination methods.

SUMMARY:
Taiwan Registry of Endovascular Thrombectomy for Acute Ischemic Stroke is a multi-centers registration. It starts in Jan 2019. The key items in the registration form include basic demographic profiles, past medical history, time of stroke onset, stroke severity (NIH stroke scale), whether to have rt-PA treatment, pre-EVT imaging, type of devices, status of recanalization, complication and other associated parameters for EVT, and 3 months post stroke outcome. The study also includes a standardized imaging analysis for the quantification of the de-identified imaging data from participates. In summary, the registry will provide the valuable information for AIS patients receiving EVT in Twain.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death and third leading cause of disability worldwide. Until recently, intravenous recombinant tissue-type plasminogen activator (r-tPA) was the only therapy that was proven to be effective for acute ischemic stroke (AIS). However, the effect of rt-PA was limited in stroke patients with large artery occlusion. In 2015, there were five randomized controlled trials of endovascular therapy (EVT) for AIS. The significant positive results indicated an evolution of treatment for AIS in selected patients. Nevertheless, because previous EVT trials recruited mainly Caucasians as trial participants, little is known about racial differences in endovascular treatment.

In Taiwan, the Ministry of Health and Welfare has approved the application of EVT in AIS and the National Health Insurance also started to pay the devices for EVT in AIS patients fulfilling certain conditions in recent years. Therefore, it is important to have a prospective registration to evaluate the efficacy and safety in AIS patients receiving EVT in Taiwan.

Taiwan Registry of Endovascular Thrombectomy for Acute Ischemic Stroke is a multi-centers registration. It starts in Jan 2019. The key items in the registration form include basic demographic profiles, past medical history, time of stroke onset, stroke severity (NIH stroke scale), whether to have rt-PA treatment, pre-EVT imaging, type of devices, status of recanalization, complication and other associated parameters for EVT, and 3 months post stroke outcome. The study also includes a standardized imaging analysis for the quantification of the de-identified imaging data from participates.

In summary, the registry will provide the valuable information for AIS patients receiving EVT in Twain.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke caused by intracranial large vessel occlusion
* Can be treated within 24 hours of stroke onset.
* Large vessel occlusion demonstrated by magnetic resonance imaging angiography (MRA), computed tomography angiography (CTA) or digital substraction angiography (DSA).
* Pre-stroke independence (modified Rankin Scale 0-2).

Exclusion Criteria:

* Other cause of stroke, such as intracranial hemorrhage.
* Not underwent endovascular thrombectomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke caused by intracranial large vessel occlusion who can be treated within 24 hours of stroke onset.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | 90 days
  Functional outcome by modified Rankin scale at 90 days post-stroke

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Chun Tang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided